CLINICAL TRIAL: NCT05026099
Title: Effects of Boxing Training on Upper Limb Function, Balance and Quality of Life in Stroke Patients
Brief Title: Boxing Training for Upper Limb Functions, Balance, and Quality of Life in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Riphah/REC/01031 Mubbra
Record Dates: First submitted 2021-08-23; First posted 2021-08-30 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Boxing training program (Experimental): The program will start with a warm-up session involving breathing and stretching of the trunk and limbs for 5 minutes. The program will include mitt hitting and sand bag hitting for 10 minutes, with a 2-minute rest period. Thereafter, stretching of the trunk and limbs will be performed for 5minutes, similar to the warm-up
  Interventions: Other: Boxing training
- Task Oriented Training Program (Active Comparator): Upper limb Exercises: Sitting position: open covered pots of different sizes and transfer the flour to a cup with a spoon, then close the pot.Sitting position: pick up coins and cards on the table and put the coins in a pot and gather the cards.Sitting position: write and/or draw pictures on a piece of paper.Sitting position: open a safe box with a key, pick up small objects inside the box, and transfer them to a pot, then lock the safe box Sitting position: pick up and transfer jars, bottles, and glasses of different sizes and weights located on a table. Transfer the liquid contents from jars and bottles to glasses Sitting position: throw and catch balls (in pairs)
  Interventions: Other: Task Oriented Training

INTERVENTIONS:
Other: Boxing training — Boxing training: warm-up. Mitt hitting, sandbag hitting, in sitting, cool down, Assessment after 4 weeks boxing training: warm-up. Mitt hitting, sandbag hitting, below hips, cool down, Assessment after 6 weeks Boxing training: warm-up. Mitt hitting, sandbag hitting, both inn sitting and standing, cool down, Post assessment
  Arms: Boxing training program
Other: Task Oriented Training — Task-oriented training: 6 tasks in sitting and standing position for both upper and lower limb Assessment after 4 weeks Task oriented training: 6 tasks in sitting and standing position for both upper and lower limb Assessment after 6 weeks Task oriented training: 6 tasks in sitting and standing position for both upper and lower limb Post assessment
  Arms: Task Oriented Training Program

SUMMARY:
The World Health Organization's (WHO) definition of stroke is a clinical syndrome characterized by rapidly developing clinical signs of focal (or global) disturbance of cerebral function lasting more than 24 hours or leading to death with no apparent cause other than a vascular origin'.Stroke has further three types i.e. ischemic, hemorrhagic, and transient ischemic stroke. As most gestures in daily life involve the upper limbs and hands, patients who cannot use their hands not only suffer from severe physical and psychological pain but also encounter difﬁculties in the activities of daily living that primarily involve upper limb function. Stroke patients have various problems such as asymmetrical posture, abnormal body balance, and decreased ability to move the weight.

DETAILED DESCRIPTION:
As most gestures in daily life involve the upper limbs and hands, patients who cannot use their hands not only suffer from severe physical and psychological pain but also encounter difﬁculties in the activities of daily living that primarily involve upper limb function. Stroke patients have various problems such as asymmetrical posture, abnormal body balance, and decreased ability to move the weight. The loss of motion element involved in ﬁne functions, and the above-mentioned problems can lead to decreased muscle cooperativity of the lower limbs while walking and may also result in an asymmetric gait due to imbalance in the ability to perform the exercise. Due to such persistent disorders, most stroke patients suffer from depression, problems in interpersonal relationships and social life, and a generally lower quality of life. Recent studies on the treatment of stroke patients reported that approaches such as more intensive and repetitive training as compared to conventional general and passive intervention, training related to reality, intervention involving motivation and active participation and forced induction exercise, visual exercise feedback, purpose-oriented training, and task-oriented training are more effective in promoting function after stroke onset. Virtual reality (VR) is frequently used in different disease groups at the clinic for rehabilitation purposes. Xbox Kinect, Nintendo Wii, Sony PlayStation, and Cyber Glove are among the most commonly used VR applications in rehabilitation. Several studies reported that VR applications improved both upper and lower extremity functions and promoted independence in performing activities of daily living. Task-specific training focused on both upper limbs and lower limbs could have a greater impact in improving mobility and physical activity in individuals with stroke but these studies have very little impact on balance, gait, and quality of life in patients with stroke. Previous studies reported that task-oriented training programs in stroke patients only focus on lower limb and upper limb function. The main barrier or limitation in task-oriented training is the repetition of tasks in an appropriate manner, and most patients lose interest and feel bored and there is less active participation during the performance of similar tasks. This will affect their performance and function and not very much effective intervention for treating stroke patients.

In recent years, it has been observed that boxing therapy has positive outcomes in individuals with neurological diseases. In the literature, the first study, including boxing therapy, was conducted in patients with Parkinson's disease, which concluded that boxing therapy was feasible and reliable for Parkinson's patients. As a form of high-intensity exercise, it is argued that goal-based activities such as boxing can be engaging and accessible for people with chronic diseases. Boxing incorporates high-intensity exercise, with movements of all regions of the body in a weight-bearing and aerobic context. Either non-contact or as a contact sport, boxing movements can be performed in sitting, standing, or as part of dynamic, complex movement sequences. In able-bodied people, high-intensity boxing programs performed for 50-minutes four times per week improved fitness, health, and well-being. The other preliminary on the effects of the sitting boxing program in stroke patients investigated and demonstrated that the sitting boxing program had a positive impact on upper extremity function, balance, gait, and quality of life in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Age 40-60years
* Middle Cerebral Artery Stroke
* Fugyl Meyer score limit for upper limb:
* Sub-acute and chronic (after 6 weeks)
* Able to sit for 2mints independently

Exclusion Criteria:

* Cognitive impairment
* Abnormal synergic pattern
* Rheumatoid arthritis or other hand impairments
* Visual Impairment

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-08-20 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment | week 8
  A three-point ordinal scale is used to measure impairments of volitional movement with grades ranging from 0 (item cannot be performed) to 2 (item can be fully performed). Specific descriptions for performance accompany individual test items. Subtests exist for Upper extremity function, Lower extremity function, balance, sensation, Range of Motion, and pain. The cumulative test score for all components is 226 with availability of specific subtest scores (e.g., Upper extremity maximum score is 66, Lower extremity score 34; balance score 14)
Wolf Motor Function Test | week 8
  the Wolf Motor Function Test consists of 17 items Composed of 3 parts:
  * Time
  * Functional ability
  * Strength Includes 15 function-based tasks and 2 strength-based tasks Performance time is referred to as Wolf Motor Function Test-Time. Functional ability is referred to as Wolf Motor Function Test. Items 1-6 involve timed functional tasks, items 7-14 are measures of strength, and the remaining 9 items consist of analyzing movement quality when completing various tasks Examiners should test the less affected upper extremity followed by the most affected side. Uses a 6-point ordinal scale "0" = "does not attempt with the involved arm" to "5" = "arm does participate; movement appears to be normal." The maximum score is 75 Lower scores are indicative of lower functioning levels Wolf Motor Function Test Time allows 120 seconds per task
Berg Balance Scale | week 8
  The maximum score that can be reached is 56 and each item possesses an ordinal scale of five alternatives ranging from 0 to 4 points.

SECONDARY OUTCOMES:
Stroke Specific Quality of life | week 8
  used to assess quality of life in stroke patients. 49 items Items are assessed on 5-point Guttman-type scales. Each item is answered using 1 of 3 different response sets.
  Provides both summary and domain specific scores:
  1. Domain scores are composed of unweighted averages
  2. Summary scores are composed of an unweighted average of the 12 domain average scores Scores range from 49-245. Higher scores indicate better functioning.
  The 12 domains include:
  1. Mobility
  2. Energy
  3. Upper Extremity Function
  4. Work and Productivity
  5. Mood
  6. Self-care
  7. Social Roles
  8. Family Roles
  9. Vision
  10. Language
  11. Thinking
  12. Personality

CONTACTS AND LOCATIONS:
Overall Officials: Arshad Malik, PhD, Principal Investigator — Riphah International University
Locations (1):
- Iradah Rehabilitation Center Kalar Kahar, Chakwal, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sacco RL, Kasner SE, Broderick JP, Caplan LR, Connors JJ, Culebras A, Elkind MS, George MG, Hamdan AD, Higashida RT, Hoh BL, Janis LS, Kase CS, Kleindorfer DO, Lee JM, Moseley ME, Peterson ED, Turan TN, Valderrama AL, Vinters HV; American Heart Association Stroke Council, Council on Cardiovascular Surgery and Anesthesia; Council on Cardiovascular Radiology and Intervention; Council on Cardiovascular and Stroke Nursing; Council on Epidemiology and Prevention; Council on Peripheral Vascular Disease; Council on Nutrition, Physical Activity and Metabolism. An updated definition of stroke for the 21st century: a statement for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2013 Jul;44(7):2064-89. doi: 10.1161/STR.0b013e318296aeca. Epub 2013 May 7. PMID 23652265
- [Background] Ersoy C, Iyigun G. Boxing training in patients with stroke causes improvement of upper extremity, balance, and cognitive functions but should it be applied as virtual or real? Top Stroke Rehabil. 2021 Mar;28(2):112-126. doi: 10.1080/10749357.2020.1783918. Epub 2020 Jun 23. PMID 32574096
- [Background] Duncan PW, Horner RD, Reker DM, Samsa GP, Hoenig H, Hamilton B, LaClair BJ, Dudley TK. Adherence to postacute rehabilitation guidelines is associated with functional recovery in stroke. Stroke. 2002 Jan;33(1):167-77. doi: 10.1161/hs0102.101014. PMID 11779907
- [Background] Park J, Gong J, Yim J. Effects of a sitting boxing program on upper limb function, balance, gait, and quality of life in stroke patients. NeuroRehabilitation. 2017;40(1):77-86. doi: 10.3233/NRE-161392. PMID 27792020
- [Background] Langhorne P, Bernhardt J, Kwakkel G. Stroke rehabilitation. Lancet. 2011 May 14;377(9778):1693-702. doi: 10.1016/S0140-6736(11)60325-5. PMID 21571152
- [Background] Kwakkel G, van Wegen EEH, Burridge JH, Winstein CJ, van Dokkum LEH, Alt Murphy M, Levin MF, Krakauer JW; ADVISORY group. Standardized Measurement of Quality of Upper Limb Movement After Stroke: Consensus-Based Core Recommendations From the Second Stroke Recovery and Rehabilitation Roundtable. Neurorehabil Neural Repair. 2019 Nov;33(11):951-958. doi: 10.1177/1545968319886477. Epub 2019 Oct 29. PMID 31660781
- [Background] Feys HM, De Weerdt WJ, Selz BE, Cox Steck GA, Spichiger R, Vereeck LE, Putman KD, Van Hoydonck GA. Effect of a therapeutic intervention for the hemiplegic upper limb in the acute phase after stroke: a single-blind, randomized, controlled multicenter trial. Stroke. 1998 Apr;29(4):785-92. doi: 10.1161/01.str.29.4.785. PMID 9550512
- [Background] Rodriguez GM, Aruin AS. The effect of shoe wedges and lifts on symmetry of stance and weight bearing in hemiparetic individuals. Arch Phys Med Rehabil. 2002 Apr;83(4):478-82. doi: 10.1053/apmr.2002.31197. PMID 11932848